CLINICAL TRIAL: NCT02422992
Title: Haptoglobin Phenotype and Smoking: Effects on Iron Levels in Parkinson's Disease
Brief Title: Haptoglobin and Iron in Parkinson's Disease
Acronym: HPPD
Status: Completed | Type: Observational
Sponsor: Bastyr University (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 12A-1330
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease
Keywords: Iron metabolism; MRI; risk factors; haptoglobin phenotype
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — We collect serum and plasma samples during the study, that were tested for total serum iron and iron-binding proteins.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PD: 100 PD patients were patients diagnosed with Parkinson's disease
- Controls: 242 Controls were subjects free of neurodegenerative diseases, matched by age and gender to the PD patients

SUMMARY:
This is a case/control epidemiology study to identify what are the iron-metabolism abnormalities in Parkinson's disease (PD) patients, and risk factors relevant to PD predisposition.

DETAILED DESCRIPTION:
A total of 342 participants, 100 PD patients and 242 age- and gender matched controls, were included in the study. All study participants were seen for one study visit in the morning at one of two Bastyr University Clinics in the Seattle area. Study participants were fasting at the time of the visit. During the study visit, participants donated a blood sample for the blood tests and complete an epidemiology questionnaire.

A subset of 51 of the study participant who were seen for the visit at Bastyr University, underwent brain scan and Magnetic Resonance Imaging (MRI), at the University of Washington Department of Radiology. The MRI part of the study aims at estimating brain iron levels.

ELIGIBILITY:
Inclusion Criteria for the Controls, for the blood draw and epidemiology visit:

* Volunteers should be of age between 52 and 82 years of age, males of females.

Exclusion Criteria for the Controls:

* presence of a neurodegenerative disease,
* presence of active cancer under treatment,
* HIV sero-positivity, Hepatitis B, C, of A sero-positivity
* rheumatoid arthritis
* recent blood donation (less than three months before the visit).
* fever at the time of the visit

Inclusion Criteria for the Parkinson's disease patients:

Diagnosis of Parkinson's disease (UKBB clinical criteria).

Exclusion criteria for the Parkinson's disease patients, for the blood draw and epidemiology visit:

* Presence of other neurodegenerative diseases, apart for Parkinson's disease
* two or more family members with Parkinson's disease
* presence of active cancer under treatment
* HIV sero-positivity, Hepatitis B, C, of A sero-positivity
* rheumatoid arthritis
* recent blood donation (less than three months before the visit).
* fever at the time of the visit

Exclusion criteria for the Magnetic Resonance Imaging:

* presence in the body of a ferro-magnetic metallic foreign object such as, but not limited to:
* a cardiac pacemaker
* aneurism clip
* neuro-stimulator
* surgical clip
* artificial limb or joint
* orthopedic items, such as screws, nails, pins, rods,
* any metallic foreign body from a previous injury, bullets, shrapnels, metal slivers.
* exclusion criteria for MRI is also the presence of claustrophobia

Ages: 35 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients will be included in the study if they received a diagnosis of Parkinson's disease that meets the United Kingdom Brain Bank (UKBB) clinical criteria of Parkinson's disease diagnosis.
  Control participants will be included in the study if free of neurodegenerative diseases.
  A subset of the study participants (60 total) receive Magnetic Resonance Imaging to estimate brain iron
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Iron metabolism differences between PD patients and controls | Up to 7 years
  Iron metabolism will be measured by testing for serum iron and iron-binding proteins, and by estimating brain iron by MRI. Serum iron parameters that will be measured include total serum iron, iron-binding proteins such as transferrin and ferritin, and tests related to iron metabolism: transferrin % saturation, unsaturated iron binding capacity, soluble transferrin receptor, complete blood count, hemoglobin, uric acid, haptoglobin, haptoglobin phenotype. Differences in serum iron parameters, and brain iron levels, between PD patients and controls will be calculated.

SECONDARY OUTCOMES:
Environmental factors affecting PD risk and gene-environment interactions | recruitment until January 2016
  Questionnaire data will be analyzed to identify risk factors for PD by comparing lifestyle and dietary patterns from questionnaire between PD cases and controls. Interaction between haptoglobin phenotype and tobacco smoking on PD risk will be calculated, as well as interaction between haptoglobin phenotype and environmental factors such as tobacco smoking and diet on serum iron and brain iron levels.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Costa-Mallen, PhD, Principal Investigator — Bastyr University
Locations (3):
- United States (3):
  - University of California, San Diego, California
  - Bastyr University Research Institute, Kenmore, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Costa-Mallen P, Checkoway H, Zabeti A, Edenfield MJ, Swanson PD, Longstreth WT Jr, Franklin GM, Smith-Weller T, Sadrzadeh SM. The functional polymorphism of the hemoglobin-binding protein haptoglobin influences susceptibility to idiopathic Parkinson's disease. Am J Med Genet B Neuropsychiatr Genet. 2008 Mar 5;147B(2):216-22. doi: 10.1002/ajmg.b.30593. PMID 17918239